CLINICAL TRIAL: NCT03226899
Title: A Phase 4, Study to Evaluate the Safety and Efficacy of Lesinurad 200 mg in Combination With a Xanthine Oxidase Inhibitor (XOI), Compared With an XOI Alone, in Subjects With Gout and Estimated Creatinine Clearance (eCrCl) 30 to <60 mL/Min Who Have Not Achieved Target Serum Uric Acid Levels (sUA) on an XOI Alone
Brief Title: A Phase 4 Safety and Efficacy Study to Evaluate Lesinurad 200 mg in Participants With Gout and Renal Impairment
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This action was a business decision & not related to any efficacy, safety or clinical concerns with lesinurad.
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-401
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Results first posted 2021-11-04 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Gout; Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Gout; Renal Insufficiency, Chronic | interventions — lesinurad; Allopurinol; Febuxostat; Colchicine; Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Multicenter, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator
Masking Description: active vs placebo visually identical tablets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lesinurad + XOI (Active Comparator): lesinurad 200 mg oral tablet QD plus a stable, medically appropriate dose of an XOI
  Interventions: Drug: Lesinurad; Drug: XOI; Drug: colchicine; Drug: corticosteroids
- Placebo + XOI (Placebo Comparator): placebo tablet QD plus a stable, medically appropriate dose of an XOI
  Interventions: Drug: XOI; Drug: Placebo; Drug: colchicine; Drug: corticosteroids

INTERVENTIONS:
Drug: Lesinurad — 200 mg oral tablet
  Other Names: RDEA594
  Arms: Lesinurad + XOI
Drug: XOI — All participants must be on a stable, medically appropriate dose of XOI as their sole urate-lowering therapy (ULT) indicated for the treatment of gout for at least 4 weeks prior to Screening and throughout the Screening Period. This stable dose of XOI will be maintained throughout the study period.
  Other Names: allopurinol; febuxostat
Drug: Placebo — matching placebo oral tablet
  Arms: Placebo + XOI
Drug: colchicine — Gout flare prophylaxis: commercially available colchicine is provided through the Month 6 study visit. Actual colchicine dose (0.5 or 0.6 mg qd) and frequency were adjusted based on the local label, subject medical history, and clinical judgement.
Drug: corticosteroids — Gout flare prophylaxis: Participants unable to take colchicine are permitted to take a short course of low-dose oral corticosteroids up to the Month 3 study visit

SUMMARY:
This study evaluates the safety and efficacy of lesinurad administered with an XOI versus a placebo plus an XOI in gout participants who have moderate renal impairment and who are not at target level of serum urate (sUA).

DETAILED DESCRIPTION:
This postmarketing study is a randomized, double-blind, placebo-controlled study to evaluate safety (with particular focus on renal and cardiovascular events) and efficacy of lesinurad 200 mg once daily (QD) in combination with an XOI for up to 24 months compared with XOI monotherapy, in participants with gout and moderate renal impairment who have not reached target sUA levels (<6.0 mg/dL) on an XOI alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is able to understand the study procedures, the risks involved, and willing to provide written informed consent before the first study related activity.
2. Subject is willing to adhere to the protocol schedule.
3. Subject is ≥ 18 years and ≤ 85 years of age.
4. Subject has a diagnosis of gout.
5. Subject has moderate renal impairment with estimated creatinine clearance (eCrCl; calculated by the Cockcroft-Gault formula using ideal body weight) 25.0 to ≤ 65.0 mL/min at Screening Visits 1 and 2 and an average eCrCl for both screening visits of 30.0 to < 60.0 mL/min.
6. Subject has been taking an XOI as ULT indicated for the treatment of gout for at least 4 weeks prior to Screening at a stable, medically appropriate dose, as determined by the Investigator. The minimum dose of allopurinol is 200 mg daily, and the minimum dose of febuxostat is the lowest approved dose per the local product label.
7. Subject has a serum uric acid level ≥ 6.0 mg/dL (357 µmol/L) at Screening Visits 1 and 2.
8. Subject is male or female; females must not be pregnant or breastfeeding and females of childbearing potential must agree to use nonhormonal contraception during the Screening Period and while taking investigation product (IP).
9. Subject has a body mass index < 45 kg/m^2.

Exclusion Criteria:

1. Subject had unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, or stroke within the last 6 months prior to randomization; or had a deep venous thrombosis within the previous 3 months prior to randomization.
2. Subject has uncontrolled hypertension (defined as systolic pressure above 160 or diastolic pressure above 95 mm Hg at either Screening Visits 1 or 2).
3. Subject has severe hepatic impairment (defined as Child-Pugh Class C) or is known human immunodeficiency virus (HIV) positive.
4. Subject is a solid organ transplant recipient.
5. Subject has a urine protein of 3+ or higher by dipstick by the central laboratory at Screening Visit 2.
6. Subject has a history of glomerulonephritis.
7. Subject is taking valpromide, progabide, valproic acid, or other known inhibitors of epoxide hydrolase, or subject is taking ranolazine, cyclosporine, azathioprine or mercaptopurine.
8. Subject is receiving chronic treatment with more than 325 mg of salicylates per day.
9. Subject is unable to initiate gout flare prophylaxis with colchicine or low-dose oral corticosteroids at Baseline.
10. Subject is taking any other drug approved for use as a urate-lowering medication other than allopurinol or febuxostat (eg, pegloticase, probenecid, benzbromarone) within 4 weeks prior to Screening or during Screening.
11. For subjects who will be taking colchicine for gout flare prophylaxis: Subject is taking, or anticipated to take during the first 6 months on study, moderate or strong Cytochrome P450 3A4 (CYP3A4) inhibitors (ie, verapamil or diltiazem, clarithromycin, and fluconazole; or grapefruit or grapefruit juice).
12. Subject previously participated in a clinical study involving lesinurad (RDEA594) or verinurad (RDEA3170) and received active treatment or placebo, or has taken commercially-available lesinurad.
13. Subject has a gout flare during the Screening Period.
14. Subject is pregnant or breastfeeding.
15. Subject consumes more than 14 drinks of alcohol per week (eg, 1 drink = 5 oz [150 mL] of wine, 12 oz [360 mL] of beer, or 1.5 oz [45 mL] of hard liquor).
16. Subject has a history of malignancy and has been on active treatment within the previous 5 years prior to randomization with the exception of non-melanoma skin cancer, treated in situ Grade 1 cervical cancer, or treated ductal carcinoma in situ of the breast.
17. Subject has been hospitalized (other than for elective surgery) or received intravenous contrast (eg, for computerized tomography (CT) scan or any angiography) within 1 month prior to Screening or during Screening.
18. Subject has participated in a clinical trial within 8 weeks prior to Screening.
19. Subject has any other medical or psychological condition, which in the opinion of the Investigator might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements or to complete the study.
20. The maximum number of subjects in the eCrCl stratification subgroup has been reached.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ironwood Study Chair, Study Chair — Ironwood Pharmaceuticals, Inc.
Locations (116):
- United States (70):
  - Central Alabama Research, Birmingham, Alabama
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Medvin Clinical Research, Covina, California
  - Northern California Research, Sacramento, California
  - Capital Nephrology Medical Group, Sacramento, California
  - Inland Rheumatology Clinical Trials, Inc, Upland, California
  - Medvin Clinical Research - Whittier, Whittier, California
  - Western Nephrology-Westminster, Westminster, Colorado
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Arthritis, Autoimmune, & Allergy LLC, Daytona Beach, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - Eastern Research, Hialeah, Florida
  - San Marcus Research Clinic Inc, Miami, Florida
  - LCC Medical Research Institute, LLC, Miami, Florida
  - Savin Medical Group, Miami Lakes, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - BayCare Medical Group, Inc., Tampa, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - The Kaufmann Clinic, Inc, Atlanta, Georgia
  - Ellipsis Group, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center PA, Idaho Falls, Idaho
  - Clinical Investigation Specialists, Inc. - Gurnee, Gurnee, Illinois
  - Nephrology Specialists, Merrillville, Indiana
  - Kansas Nephrology Research Institute, Wichita, Kansas
  - Center for Arthritis & Osteoporosis, Elizabethtown, Kentucky
  - Four Rivers Clinical Research, Paducah, Kentucky
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Clinical Trials Management, LLC - Northshore, Covington, Louisiana
  - Clinical Trials Management LLC - Southshore, Metairie, Louisiana
  - Arthritis and Diabetes Clinic, Monroe, Louisiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Kidney Consultants, Pontiac, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - CRC of Jackson, LLC, Jackson, Mississippi
  - VA Medical Center - Kansas City, Kansas City, Missouri
  - Meridian Clinical Research - Norfolk, NE, Norfolk, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center Inc., Albuquerque, New Mexico
  - Ellipsis Research Group, LLC, Brooklyn, New York
  - Buffalo VA Medical Center, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - DJL Clinical Research PLLC, Charlotte, North Carolina
  - PhysiqueMed Clinical Trials, Greensboro, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Sterling Research Group, Ltd. - Auburn, Cincinnati, Ohio
  - Sterling Research Group, Ltd. - Cincinnati, Cincinnati, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Columbia Research Group, Inc., Portland, Oregon
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, East Providence, Rhode Island
  - Low Country Rheumatology, Charleston, South Carolina
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - Mountain View Clinical Research - Greer, Greer, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Discovery Alliance International Inc. d/b/a Tennessee Health Research Alliance LLC, Nashville, Tennessee
  - Nephrology Associates, P.C., Nashville, Tennessee
  - FMC Science, Lampasas, Texas
  - P&I Clinical Research, Lufkin, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Briggs Clinical Research, Inc., San Antonio, Texas
  - 3rd Coast Research Associates, Victoria, Texas
  - Spectrum Medical, Inc., Danville, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
- Czechia (11):
  - CCBR Czech Brno, s. r. o, Brno
  - REVMACLINIC s.r.o. - Revmatologicka ambulance, Brno
  - DTTO Faculty Hospital Brno, Brno
  - Revmatologie MUDr. Bilkova s.r.o., Olomouc
  - CCBR Ostrava s.r.o., Ostrava
  - CCBR Clinical Research, Pardubice, Pardubice
  - CCBR Czech Prague s.r.o., Prague
  - MEDICAL PLUS, s.r.o. - Revmatologicka ambulance, Uherské Hradiště
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem
  - PV - MEDICAL, s.r.o., Zlín
  - Nemocnice Znojmo p.o - Interni oddeleni, Znojmo
- Hungary (13):
  - Bajai Szent Rokus Korhaz, Baja
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Dr Lakatos Ferenc Belgyogyaszati-Kardiologiai Maganrendelo, Békéscsaba
  - Clinexpert Kft., Budapest
  - Vaszary Kolos Korhaz Esztergom - Reumatologiai osztaly, Esztergom
  - BKS Research Kft., Hatvan
  - Kalocsai Szent Kereszt Korhaz, Kalocsa
  - Selye Janos Hospital - Rheumatology Department, Komárom
  - CRU Hungary Kft., Miskolc
  - Clinfan Ltd SMO, Szekszárd
  - Mentahaz Maganorvosi Kozpont (SMO), Székesfehérvár
  - Allergo-Derm Bakos Kft., Szolnok
  - Medical Expert Kft., Veszprém
- Poland (22):
  - Stacja Dializ Zyrardow, Żyrardów, Zyrardo
  - B_Serwis Popenda Sp. J., Chorzów
  - Centrum Kliniczno Badawcze J. Brzezicki B. Gornikiewicz - Brzezicka Lekarze Sp. p., Elblag
  - MCBK s.c., Grodzisk Mazowiecki
  - NZOZ Praktyka Lekarza Rodzinnego Elzbieta Kelm, Katowice
  - Centrum Medyczne Pratia Krakow, Krakow
  - Malopolskie Centrum Medyczne, Krakow
  - Samodzielny Publiczny ZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Oddzial Kliniczny Nefrologii, Hipertensjologii i Transplantologii Nerek, Lodz
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo Akcyjna, Lodz
  - AppleTreeClinics Sp. z o.o., Lodz
  - Centrum Medyczne AMED Oddzial w Lodzi, Lodz
  - NZOZ All - Med Centrum Medyczne Specjalistyczne Gabinety Lekarskie Marcin Ogorek, Lodz
  - Centrum Medyczne Chodzki, Lublin
  - Alfa Specjalistyczne Gabinety Lekarskie Ewa Moroz, Nowy Sącz
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Centrum Badan Klinicznych s.c., Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Prywatny Gabinet Lekarski NZOZ Centrum Medyczne Aeskulap, Radom
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - KO - MED Centra Kliniczne Sp. z o.o., Osrodek Badan Klinicznych w Zamosciu, Zamość
  - Centrum Dializa Sp. z o.o. - Zyrardow, Żyrardów

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo + XOI: Placebo oral tablet once daily (QD) plus a stable, medically appropriate dose of an xanthine oxidase inhibitor (XOI)
Period: Overall Study
Arm/Group | Placebo + XOI | Lesinurad + XOI
Started | 118 | 124
Completed (completed the study/24 months of treatment) | 0 | 0
Not Completed | 118 | 124

BASELINE CHARACTERISTICS:
Groups:
- Placebo + XOI: placebo oral tablet QD plus a stable, medically appropriate dose of an XOI
- Total: Total of all reporting groups
Arm/Group | Placebo + XOI | Lesinurad + XOI | Total
Number analyzed (Participants) | 118 | 124 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (8.00) | 66.4 (10.10) | 66.8 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 96 | 96 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 20 | 46
  Not Hispanic or Latino | 92 | 104 | 196
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 14 | 24 | 38
  White | 99 | 95 | 194
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Serum Urate (sUA) < 6.0 mg/dL at Month 6
Time Frame: Month 6
Population: Modified Intent-to-Treat (mITT) Population: all randomized participants who received at least 1 dose of study drug. Participants with a value at Month 6.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 80 | 80
percentage of participants | 33.8 | 58.8

2. Secondary Outcome: Percentage of Participants Who Achieve sUA < 6.0 mg/dL Over Time
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18
Population: mITT Population: all randomized participants who received at least 1 dose of study drug. Participants with a value at baseline and given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
percentage of participants
  Baseline | 10.3 | 10.6
  Month 1: number analyzed (Participants) | 111 | 119
  Month 1 | 35.1 | 58.8
  Month 3: number analyzed (Participants) | 99 | 101
  Month 3 | 36.4 | 52.5
  Month 6: number analyzed (Participants) | 80 | 80
  Month 6 | 33.8 | 58.8
  Month 9: number analyzed (Participants) | 50 | 42
  Month 9 | 34.0 | 42.9
  Month 12: number analyzed (Participants) | 28 | 23
  Month 12 | 42.9 | 56.5
  Month 15: number analyzed (Participants) | 11 | 8
  Month 15 | 45.5 | 62.5
  Month 18: number analyzed (Participants) | 1 | 0
  Month 18 | 0.0 |

3. Secondary Outcome: Change From Baseline in sUA Over Time, Including the Last Value On and Off Treatment
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18
Population: Safety Population: all randomized participants who received at least 1 dose of lesinurad or placebo. Participants with a value at baseline and given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
µmol/L
  Change at Month 1: number analyzed (Participants) | 111 | 119
  Change at Month 1 | -57.0 (96.2) | -120.3 (105.3)
  Change at Month 3: number analyzed (Participants) | 99 | 101
  Change at Month 3 | -59.8 (98.6) | -106.8 (116.2)
  Change at Month 6: number analyzed (Participants) | 80 | 80
  Change at Month 6 | -54.6 (103.1) | -125.8 (140.0)
  Change at Month 9: number analyzed (Participants) | 50 | 42
  Change at Month 9 | -70.6 (128.4) | -95.9 (106.5)
  Change at Month 12: number analyzed (Participants) | 28 | 23
  Change at Month 12 | -78.7 (122.4) | -69.6 (110.4)
  Change at Month 15: number analyzed (Participants) | 11 | 8
  Change at Month 15 | -92.6 (91.4) | -116.6 (76.3)
  Change at Month 18: number analyzed (Participants) | 1 | 0
  Change at Month 18 | 0.00 (NA) — 1 participant at this time point. |
  Change at Last On-Treatment Visit: number analyzed (Participants) | 111 | 119
  Change at Last On-Treatment Visit | -57.0 (104.7) | -125.5 (121.4)
  Change at Last Off-Treatment Visit: number analyzed (Participants) | 6 | 11
  Change at Last Off-Treatment Visit | -70.7 (105.4) | -156.6 (149.2)

4. Secondary Outcome: Percent Change From Baseline in sUA Over Time, Including the Last Value On and Off Treatment
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
percent change
  Change at Month 1: number analyzed (Participants) | 111 | 119
  Change at Month 1 | -11.3 (18.8) | -24.0 (19.3)
  Change at Month 3: number analyzed (Participants) | 99 | 101
  Change at Month 3 | -11.4 (18.8) | -21.2 (21.7)
  Change at Month 6: number analyzed (Participants) | 80 | 80
  Change at Month 6 | -10.0 (21.7) | -23.9 (24.4)
  Change at Month 9: number analyzed (Participants) | 50 | 42
  Change at Month 9 | -12.6 (27.3) | -18.6 (20.2)
  Change at Month 12: number analyzed (Participants) | 28 | 23
  Change at Month 12 | -15.2 (22.8) | -14.7 (26.7)
  Change at Month 15: number analyzed (Participants) | 11 | 8
  Change at Month 15 | -18.9 (17.5) | -26.1 (16.3)
  Change at Month 18: number analyzed (Participants) | 1 | 0
  Change at Month 18 | 0.00 (NA) — 1 participant at this time point. |
  Change at Last On-Treatment Visit: number analyzed (Participants) | 111 | 119
  Change at Last On-Treatment Visit | -10.6 (22.1) | -24.8 (22.8)
  Change at Last Off-Treatment Visit: number analyzed (Participants) | 6 | 11
  Change at Last Off-Treatment Visit | -16.1 (25.8) | -27.3 (22.6)

5. Secondary Outcome: Change From Baseline in Estimated Creatinine Clearance (eCrCl) at Month 24
Description: The eCrCl was calculated by the Cockcroft-Gault formula using ideal body weight.
Time Frame: Baseline, 24 months
Population: Due to early study termination, no participant reached Month 24. Therefore these data are not available.
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percent Change From Baseline in eCrCl at Month 24
Description: The eCrCl was calculated by the Cockcroft-Gault formula using ideal body weight.
Time Frame: Baseline, 24 months
Population: Due to early study termination, no participant reached Month 24. Therefore these data are not available.
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change From Baseline in eCrCl Over the Study Period, Including the Last Value On and Off Treatment
Description: The eCrCl was calculated by the Cockcroft-Gault formula using ideal body weight.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
mL/min
  Change at Month 1: number analyzed (Participants) | 111 | 119
  Change at Month 1 | 0.13 (9.67) | -1.29 (6.45)
  Change at Month 3: number analyzed (Participants) | 99 | 101
  Change at Month 3 | -0.69 (7.41) | -1.53 (8.65)
  Change at Month 6: number analyzed (Participants) | 80 | 80
  Change at Month 6 | -1.84 (7.58) | -1.80 (7.02)
  Change at Month 9: number analyzed (Participants) | 50 | 42
  Change at Month 9 | -0.78 (6.85) | -2.10 (7.97)
  Change at Month 12: number analyzed (Participants) | 28 | 23
  Change at Month 12 | -2.14 (7.03) | -4.30 (6.34)
  Change at Month 15: number analyzed (Participants) | 11 | 8
  Change at Month 15 | 0.36 (6.07) | -6.00 (8.49)
  Change at Month 18: number analyzed (Participants) | 1 | 0
  Change at Month 18 | -19.0 (NA) — 1 participant at this time point. |
  Change at Last On-Treatment Visit: number analyzed (Participants) | 111 | 119
  Change at Last On-Treatment Visit | -1.03 (6.97) | -1.91 (8.19)
  Change at Last Off-Treatment Visit: number analyzed (Participants) | 6 | 11
  Change at Last Off-Treatment Visit | 2.33 (5.61) | -2.45 (5.41)

8. Secondary Outcome: Percent Change From Baseline in eCrCl Over the Study Period, Including the Last Value On and Off Treatment
Description: The eCrCl was calculated by the Cockcroft-Gault formula using ideal body weight.
Time Frame: Baseline, Months 1, 3, 6, 9, 12, 15, 18
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
percent change
  Change at Month 1: number analyzed (Participants) | 111 | 119
  Change at Month 1 | 1.16 (19.90) | -2.07 (15.30)
  Change at Month 3: number analyzed (Participants) | 99 | 101
  Change at Month 3 | -0.18 (17.70) | -2.14 (20.12)
  Change at Month 6: number analyzed (Participants) | 80 | 80
  Change at Month 6 | -2.49 (17.96) | -3.01 (15.32)
  Change at Month 9: number analyzed (Participants) | 50 | 42
  Change at Month 9 | -0.26 (18.67) | -3.42 (17.05)
  Change at Month 12: number analyzed (Participants) | 28 | 23
  Change at Month 12 | -3.38 (15.71) | -8.1 (12.9)
  Change at Month 15: number analyzed (Participants) | 11 | 8
  Change at Month 15 | 3.67 (18.6) | -11.0 (16.5)
  Change at Month 18: number analyzed (Participants) | 1 | 0
  Change at Month 18 | -31.7 (NA) — 1 participant at this time point. |
  Change at Last On-Treatment Visit: number analyzed (Participants) | 111 | 119
  Change at Last On-Treatment Visit | -1.13 (16.86) | -3.04 (18.21)
  Change at Last Off-Treatment Visit: number analyzed (Participants) | 6 | 11
  Change at Last Off-Treatment Visit | 4.14 (13.67) | -5.35 (13.52)

9. Secondary Outcome: Percentage of Participants With Serum Creatinine (sCr) Elevations (≥1.5 × Baseline) Over the Study Period
Time Frame: up to 18 months
Population: Safety Population: all randomized participants who received at least 1 dose of lesinurad or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
percentage of participants | 5.2 | 7.3

10. Secondary Outcome: Percentage of Participants Meeting Criteria (eg, Based on sCr or eCrCl Criteria) for Treatment Discontinuations Over the Study Period
Description: Kidney function was monitored throughout the study by measuring sCr and calculating eCrCl by Cockcroft-Gault formula using ideal body weight. Treatment discontinuations were required if a participant experienced an absolute sCr ≥4.0 mg/dL or an eCrCl <20 mL/min (based on central laboratory results).
Time Frame: up to 18 months
Population: Safety Population: all randomized participants who received at least 1 dose of lesinurad or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 116 | 123
percentage of participants | 0.0 | 0.0

11. Secondary Outcome: Percentage of Participants Renal-Related and Kidney Stone Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Renal-related and kidney stone events were based on Medical Dictionary for Regulatory Activities (MedDRA) "Renal and Urinary Disorders" system organ classification. AEs that started on or after the first dose of study drug in this study, or those AEs with onset prior to the first dose of study drug but worsened after the first dose of study drug, were considered treatment emergent.
Time Frame: From first dose of study drug through each participant's study duration, up to approximately 18 months.
Population: All Randomized Participants
Measure: Number; unit: percentage of participants
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 118 | 124
percentage of participants
  Treatment-Emergent SAEs | 0.0 | 0.8
  Treatment-Emergent AEs | 4.2 | 5.6

12. Secondary Outcome: Percentage of Participants With Contributing Factors to Renal SAEs as Adjudicated by the Renal Event Adjudication Committee (REAC)
Time Frame: From first dose of study drug through each participant's study duration, up to approximately 18 months.
Population: This was not analyzed; no events were adjudicated since the study was terminated early.
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Participants With Cardiac Event Adjudication Committee (CEAC)-Adjudicated Major Adverse Cardiovascular Events (MACEs)
Description: MACEs are defined as Cardiovascular Death, Nonfatal Myocardial Infarction, and Nonfatal Stroke.
Time Frame: From first dose of study drug through each participant's study duration, up to approximately 18 months.
Population: This was not analyzed; no events were adjudicated since the study was terminated early.
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Incidence of CEAC-Adjudicated MACEs or Hospitalization for Unstable Angina (MACE+)
Description: MACEs are defined as Cardiovascular Death, Nonfatal Myocardial Infarction, and Nonfatal Stroke.
Time Frame: From first dose of study drug through each participant's study duration, up to approximately 18 months.
Population: This was not analyzed; no events were adjudicated since the study was terminated early.
Arm/Group | Placebo + XOI | Lesinurad + XOI
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug through each participant's study duration, up to approximately 18 months.
Arm/Group | Placebo + XOI | Lesinurad + XOI
All-Cause Mortality (participants affected / at risk) | 0/118 | 0/124
Serious Adverse Events (participants affected / at risk) | 7/118 | 13/124
Other Adverse Events (participants affected / at risk) | 9/118 | 18/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + XOI (N=118) | Lesinurad + XOI (N=124)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Vascular stent occlusion (General disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + XOI (N=118) | Lesinurad + XOI (N=124)
Viral upper respiratory tract infection (Infections and infestations) | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Hypertension (Vascular disorders) | 4 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may publish or disclose the results of the study 24 months after final data lock provided that sponsor can review the publication prior to public release, sponsor can request removal of confidential information of sponsor (not including results of trial), and sponsor can request a publication delay in order to protect potentially patentable information. Furthermore, if a publication committee is developing an initial publication, PI is to delay disclosure until that publication is published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT03226899/Prot_SAP_000.pdf